CLINICAL TRIAL: NCT05432414
Title: Pomalidomide, Bortezomib and Dexamethasone (PVd) Versus Bortezomib and Dexamethasone (Vd) in NDMM Patients With Renal Injury (RI)：A Multicenter, Randomized Controlled, Open-label Trial.
Brief Title: PVd Versus Vd in NDMM Patients With RI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Peking University People's Hospital (Other); Shanghai Changzheng Hospital (Other); Shanghai 6th People's Hospital (Other); Peking University Shenzhen Hospital (Other); The Third People's Hospital of Chengdu (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Ningbo No. 1 Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POM-MM-003
Record Dates: First submitted 2022-06-06; First posted 2022-06-27 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma
Keywords: NDMM with RI
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: 2(PVD):1(VD) random inclusion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pomalidomide, Bortezomib and Dexamethasone (PVD) (Experimental): Each cycle is 21 days, after 2 cycles, patients who reached MR continued treatment for 2 cycles, 4 cycles in total. Subsequent treatment regimens after 4 cycles of induction therapy were determined by the investigator.
  Interventions: Drug: pomalidomide; Drug: Bortezomib; Drug: Dexamethasone
- Bortezomib and Dexamethasone (VD) (Active Comparator): Each cycle is 21 days, after 2 cycles, patients who reached MR continued treatment for 2 cycles, 4 cycles in total. Subsequent treatment regimens after 4 cycles of induction therapy were determined by the investigator.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: pomalidomide — Pomalidomide was administered orally at a dose of 4 mg on days 1-14 of each cycle.
  Other Names: CC-4047
  Arms: Pomalidomide, Bortezomib and Dexamethasone (PVD)
Drug: Bortezomib — Bortezomib was administered intravenously or subcutaneously at a dose of 1.3mg/m2 on days 1, 4, 8, 11 of each cycle.
Drug: Dexamethasone — Dexamethasone was administered orally at a dose of 20mg on days the same and next day of bortezomib administration.

SUMMARY:
This is a multicenter, randomized controlled, open-label study, and the purpose of this study is to compare the efficiency and safety of PVD regimen (Pomalidomide & Bortezomib & Dexamethasone) versus VD regimen (Bortezomib & Dexamethasone) in NDMM patients with RI. The main efficacy indicator is VGPR after 4 cycles of induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of symptomatic multiple myeloma (according to the International Myeloma Working Group [IMWG] diagnostic criteria)
* Men and women aged ≥18 years and ≤75 years
* Multiple myeloma patients with measurable M protein should meet at least one of the following three tests: 1) Serum M protein ≥10 g/L; 2) Urinary M protein ≥200 mg/24h; 3) In the case of abnormal serum free light chain ratio, the level of affected free light chain ≥100 mg/L
* No prior treatment for multiple myeloma
* ECOG score ≤2, and predicted survival ≥3 months
* Clinically diagnosed multiple myeloma-related renal injury with calculated or measured creatinine clearance (CrCl)≥15 mL/min and < 60 mL/min (excluding patients undergoing dialysis). The calculated CrCl should be calculated using the widely accepted formula (i.e. Cockcroft-gault formula) :([140-Age] × body weight [kg] / [72 × creatinine mg/dL]); If the subject is female, multiply the result by 0.85 (1mg/dL=88.4umol/L)
* Hematology: When myeloma cells < 50%, ANC≥1.0×109/L (including with g-CSF support) and PLT≥75×109/L; Myeloma cells ≥50%, any ANC and PLT≥30×109/L; Adjusted serum calcium level ≤3.4 mmol/L; Hemoglobin level ≥8 g/dL
* For the use of symptomatic and supportive therapy only, the biochemical requirements of 6 and 7 achieved by non-myeloma treatment drugs can also be included in the group
* Liver, heart and other major organs meet the requirements of the following laboratory examination indicators (conducted within 7 days before treatment): 1) Total bilirubin ≤ 1.5 times the upper limit of normal value (same age); 2) Aspartate aminotransferase (AST) and alanine transferine (ALT) ≤ 1.5 times the upper limit of normal value (same age); 3) myocardial enzymes < 2 times the upper limit of normal value; 4) Echocardiography (ECHO) determined that cardiac ejection fraction was within the normal range.
* Patients with inactive hepatitis and total bilirubin, AST and ALT meeting the inclusion criteria, but HBV-DNA≥104, are recommended to be treated with entecavir and other antiviral drugs, and the treatment course will be determined by researchers after their own evaluation of the patient's situation
* Women of reproductive age (FCBP) subjects must have a negative serum pregnancy test 21 days prior to enrollment and consent to use a valid contraceptive method during all study medications and within 30 days after the last study medication (pregnancy tests may be performed more frequently if local guidelines are followed). FCBP is defined in this protocol as sexually mature women who: 1) have not undergone hysterectomy, bilateral oophorectomy or bilateral salpingectomy, or 2) have not experienced spontaneous menopause for at least 24 consecutive months (i.e., have had menstruation at any time in the previous 24 consecutive months)
* If having sex with FCBP, male subjects must use an effective barrier method of contraception during the study period and for 3 months after the last study drug. Male subjects were not allowed to donate sperm during treatment and for 90 days after the last study drug. Male subjects whose partners are pregnant must abstain from sex or use condoms during vaginal intercourse
* Clearly understand the test content, voluntarily participate in and complete the test, and sign the informed consent. Informed consent was signed by the patient himself or his immediate family. Considering the patient's condition, if the patient's signature is not conducive to treatment, the informed consent shall be signed by the legal guardian or the patient's immediate family member
* Those who can receive and use antithrombotic drugs, such as low-molecular-weight heparin sodium or aspirin, etc.

Exclusion Criteria:

* Primary renal disease or secondary renal injury not related to multiple myeloma, such as diabetes
* Prior treatment for myeloma (excluding radiation, bisphosphonates, or a single short-term hormone therapy [i.e., a 4-day dose less than or equivalent to dexamethasone 40mg/ day])
* Non-active multiple myeloma, including MGUS and smoking myeloma
* Prior malignancies requiring treatment or with evidence of recurrence in the 5 years prior to the first study [excluding basal cell carcinoma of the skin and the following carcinomas in situ: Squamous cell carcinoma, carcinoma in situ of bladder, carcinoma in situ of endometrium, carcinoma in situ of cervix/dysplasia, occasional histological discovery of prostate cancer (TNM stage T1a or T1b) or carcinoma in situ of breast]
* Patients with renal insufficiency accompanied by dialysis (excluding those who had received dialysis treatment due to renal insufficiency in the early stage but had not received anti-MM treatment and were not on dialysis at the time of enrollment)
* Active hepatitis A, B, C infection or known HCV RNA positive
* Known to be HIV positive
* Active infections that are not under control
* History of VTE or cerebral infarction before treatment
* Patients had uncontrolled or severe cardiovascular disease, including myocardial infarction within 6 months prior to enrollment, NYHA defined class ⅲ - ⅳ heart failure, uncontrolled angina, congestive heart failure, clinically significant pericardial disease, or cardiac amyloidosis (NT-Pro-BNP≥1800pg/mL)
* Patients who received major operations within 30 days before the enrollment, which would cause significant physical decline and increased risk of thrombosis, or the operations were scheduled during the study period. Participants who planned to undergo surgery under local anesthesia that would not significantly affect the patient's physical performance or significantly increase the risk of thrombosis could participate in the study
* The proportion of peripheral plasma cells ≥5%, and/or the absolute value of peripheral plasma cells ≥0.5×109/L
* Subjects are pregnant or lactating women
* Uncontrolled high blood pressure or uncontrolled diabetes
* Allergic to borate, mannose, and thalidomide
* According to the protocol or the investigator's judgment, the patient's serious physical or mental illness may interfere with the clinical study participation; Substance abuse, medical, psychological, or social conditions that may interfere with subjects' participation in the study or evaluation of study results
* Patients receiving other experimental drugs
* Participants in other clinical trials within one month
* Any patients deemed unsuitable for inclusion by other investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
≥very good partial response | At end of cycle 4 (each cycle is 21 days)
  The sum of a complete response and a very good partial response

SECONDARY OUTCOMES:
MRD negative rate | From randomization to the date of first documented evidence of PD until study completion, an average of 1.5 year
  When patients reached CR, NGF was used to detect the proportion of patients with bone marrow clonoplasma cells without phenotypic abnormalities. The minimum detection sensitivity was 1 clonoplasma cell in 10000 nucleated cells
immunologic function | At day 1±3 of cycle 2-5 (each cycle is 21 days)
  Twelve cytokine assays, lymphocyte subsets and absolute count, Treg cell assays, lymphocyte activation marker assays, TH1/TH2/TH17 subsets of cytokines assays
renal tubular function | At day 1±3 of cycle 2-5 (each cycle is 21 days)
  Renal remission rate was evaluated according to the 2016 IMWG expert consensus on MM renal injury
safety（Number of adverse events ） | Each cycle (each cycle is 21 days), up to 24 months of follow-up
  Number of adverse events according to symptoms, physical examination and scheduled laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Jian Hou, PhD, Principal Investigator — RenJi Hospital
Locations (1):
- Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No